CLINICAL TRIAL: NCT00289510
Title: Single-Blind, Randomized, Controlled Phase I/II Study to Compare the Safety and Immunogenicity of an Inactivated Influenza Vaccine (Whole Virion, Vero Cell Derived) With a License Egg Derived Influenza Vaccine
Brief Title: Safety and Immunogenicity Study of an Inactivated Influenza Vaccine (Whole Virion, Vero Cell Derived)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 710501
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2007-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Inactivated influenza vaccine (whole virion, Vero cell-derived)
Biological: Inactivated influenza vaccine (egg derived) [licensed control vaccine]

SUMMARY:
The objective of this study is to assess the safety and immunogenicity of inactivated influenza vaccine (whole virion, Vero cell derived). Subjects will be randomly assigned to receive a single injection of whole virion, Vero cell derived or egg derived influenza vaccine on Day 0. Subjects will return to the study site for safety evaluation at predetermined intervals for 180 days after vaccination. Subjects will also have blood drawn at predetermined intervals to measure their immunologic response to vaccination.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects who

* are 18 to 45 years of age, inclusive, on the day of screening;
* have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry;
* are clinically healthy (in a physical condition such that the physician would have no reservations vaccinating with an influenza vaccine outside the scope of a clinical study);
* agree to keep a daily record of symptoms;
* if female and capable of bearing children - have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Subjects who

* have received any influenza vaccination for the 2005/2006 influenza season and/or the 2004/2005 influenza season;
* have received any vaccination within 2 weeks prior to vaccination in this study;
* suffer from any kind of immunodeficiency;
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immune response;
* have a history of inflammatory or degenerative neurological disease (e.g. Guillain Barré, multiple sclerosis);
* have received a blood transfusion or immunoglobulins within 30 days of study entry;
* have donated blood or plasma within 30 days of study entry;
* have a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to eggs, allergy to components of the test or comparator vaccine, other known contraindications);
* have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating;
* have a known or suspected problem with alcohol or drug abuse;
* are unable to lead an independent life as a result of either physical or mental handicap;
* were administered an investigational drug within six weeks prior to study entry;
* are concurrently participating in a clinical study that includes the administration of an investigational product;
* if female, are pregnant or lactating;
* are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 423
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Markus Müller, MD, Principal Investigator — Allgemeines Krankenhaus Wien (General Hospital Vienna); Kasra Shakeri-Nejad, MD, Principal Investigator — Klinikum Westend, Berlin; Bernhard Schmitt, MD, Principal Investigator — Internistische Gemeinschaftspraxis (Group practice for internal medicine) Dr. Regner & Dr. Schmitt, Mainz; Alen Jambrecina, MD, Principal Investigator — MDS Pharma Services Germany GmbH, Hamburg; Stephan De la Motte, MD, Principal Investigator — Harrison Clinical Research / Clinical Unit, Munich
Locations (3):
- Allgemeines Krankenhaus Wien (General Hospital Vienna), Vienna, Austria
- Germany (2):
  - Klinikum Westend, Haus 18, Berlin
  - Internistische Gemeinschaftspraxis Dr. Regner & Dr. Schmitt (Group practice for internal medicine), Mainz